CLINICAL TRIAL: NCT06015529
Title: Diagnostic Strategy for Suspected Pulmonary Embolism in Emergency Departments Based on the 4-Level Pulmonary Embolism Clinical Probability Score: SPEED&PEPS Trial
Brief Title: Diagnostic Strategy for Suspected Pulmonary Embolism Based on 4PEPS
Acronym: SPEED&PEPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 36553108
Record Dates: First submitted 2023-07-31; First posted 2023-08-29 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism; suspected PE; diagnostic strategy; clinical probability; cluster-randomized trial
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Pragmatic cluster-randomized trial
Masking Description: blinded adjudication committee assessing endpoints
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group - current practices (No Intervention): The investigating physicians of the participating centers in the control group will be free to provide care as they see fit. However, a reminder of national and European guidelines for PE management will be given to them and they will have the recommendation to apply a validated strategy. To make it easier, the different scores will be included in the clinical help-decision support software called SPEED. Investigators will be asked to enter data about the included patients directly into SPEED, which will act as the study's electronic case report form (eCRF). A paper version of the CRF will also be available.
- Intervention group - 4PEPS strategy (Active Comparator): Physicians of the participating centers in the intervention group will have the recommendation to apply the 4PEPS strategy. To make it easier to apply, the 4PEPS score will be included in SPEED. Investigators will be asked to enter the information relating to patients included in the study directly into SPEED before performing any testing. Entering these data will enable the 4PEPS score to be calculated automatically and specific recommendations to be provided. A paper version of the CRF will also be available
  Interventions: Diagnostic Test: 4PEPS strategy

INTERVENTIONS:
Diagnostic Test: 4PEPS strategy — Physicians of the participating centers in the intervention group will have the recommendation to apply the 4PEPS strategy. Using 12 variables, 4PEPS defines four levels of CP that rule out a PE, namely
  1. based only on clinical data (very low CP: PEPS < 0),
  2. based on a D-dimer level < 1000 μg/L (low CP: PEPS ≥ 0 and < 5),
  3. based on a D-dimer level with an age-adjusted cut-off value (moderate CP: PEPS ≥ 5 and <12), or
  4. the diagnosis cannot reliably be ruled out based on a D-dimer test (high CP: PEPS ≥ 12)
  Arms: Intervention group - 4PEPS strategy

SUMMARY:
The increased use of diagnostic imaging and especially computed tomography pulmonary angiography in patients suspected of pulmonary embolism (PE) is an important point of concerns.

The goal of this pragmatic cluster-randomized trial is to compare the diagnostic strategy based on the four-level pulmonary embolism probability score (4PEPS) and current practices.

The main questions it aims to answer is: "Does the diagnostic strategy based on 4PEPS significantly reduce the use of thoracic imaging without increasing the risk of serious adverse events as compared to current diagnostic practices?" Patients suspected of having PE in the participating emergency departments will be included and followed for 90 days. In ten centers, the emergency physicians will apply the 4PEPS strategy and in ten other centers, the emergency physicians will be free to do as they see fit. Researchers will compare the two groups of patients to see if the rate of diagnostic thoracic imaging tests and the rate of adverse events related to diagnostic strategies will differ.

DETAILED DESCRIPTION:
Several strategies have been devised to safely limit the use of thoracic imaging in patients suspected of pulmonary embolism (PE). However, they are based on different rules for clinical probability (CP) assessment, rendering their combination difficult. The four-level pulmonary embolism probability score (4PEPS) allows the combination of all other strategies using a single CP assessment. Methods and analysis: SPEED&PEPS is a pragmatic cluster-randomized trial. After a preliminary period aimed to assess the possibility of inclusions and current practices in 23 Emergency Departments (ED), 20 EDs will be selected to participate to the active phase and randomization. Half of the centers will be allocated to the control group where physicians will be free to do as they see fit but they will be given the recommendation to apply a validated strategy. Half of the centers will be allocated to the interventional group where the physicians will be given the recommendation to apply the 4PEPS strategy. Patients with suspected PE will be included and followed for 90 days (anticipated number of patients to be included: 2560, 1280 in each arm). The primary objective will be to demonstrate that the application of the 4PEPS strategy by emergency physicians, in comparison to current practices, (i) does not increase the risk of serious events related to diagnostic strategies and (ii) significantly reduces the use of thoracic imaging. If successful, the SPEED&PEPS trial will have an important impact for patients suspected of PE limiting their irradiation and for public health in substantial savings in terms of the direct cost of diagnostic investigations and the indirect cost of hospitalizations due to waiting times or delayed harmful effects. Funding: This work is funded by a French Public Health grant (PREPS-N 2019). The funding source plays no role in the study design, data collection, analysis, interpretation or the writing of the manuscript.

ELIGIBILITY:
Inclusion Criteria:

* Admission to an emergency department participating in the study.
* Suspected PE due to thoracic symptoms (dyspnea, chest pain, or hemoptysis) and/or syncope without any other obvious explanation after clinical examination and possible additional first-line tests (ECG, chest X-ray, or routine lab work-up).

Exclusion Criteria:

* Age < 18 years.
* Known result of a specific diagnostic imaging examination for PE (thoracic CT angiography, pulmonary scintigraphy, or venous ultrasound of the lower limbs).
* Hemodynamic instability (systolic blood pressure < 90 mmHg or more than 40 mmHg lower than usual for more than 15 min).
* Curative dose of anticoagulant in place for more than two days prior to inclusion.
* Pregnant or parturient patient.
* Patient in detention by judicial or administrative decision.
* Patient undergoing compulsory psychiatric treatment.
* Patient placed under a legal protection measure.
* Patient who objects to participating in the research (preliminary phase) or is unable to give free and informed consent (active phase).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2951 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Rate of serious clinical events in the 90 days following inclusion | 90 days
  The primary safety endpoint will be the rate of serious clinical events in the 90 days following inclusion: • Serious adverse events related to diagnostic testing (leading to hospitalization or prolongation of hospitalization, permanent inability or incapacity, and death). • Symptomatic thromboembolic events in patients not diagnosed with PE in the emergency department or new thromboembolic events in patients diagnosed with PE. • Death related to PE (initial or recurrent PE). • Major bleeding related to an anticoagulant treatment prescribed for pulmonary embolism according to ISTH criteria.
Rate of diagnostic thoracic imaging | up to 72 hours following inclusion
  The primary efficacy endpoint will be the rate of thoracic imaging among all included patients with suspected PE. The following examinations are considered if they are performed at the request of the emergency physician in search of PE: computed tomography pulmonary angiography (CTPA), planar perfusion or perfusion-ventilation scintigraphy, and SPECT scintigraphy.

SECONDARY OUTCOMES:
Rate of thromboembolic events occurring in the 90 days following inclusion in patients for whom PE was ruled out according to the 4PEPS strategy in the intervention group | 90 days
  The first secondary objective is to demonstrate, in the intervention group, that the risk of false-negative diagnosis with the 4PEPS strategy is very low in accordance with the International Society of Thrombosis and Hemostasis (ISTH) criteria for validation of rule-out PE diagnostic strategies.
  The endpoint will be the false-negative rate defined as the rate of thromboembolic events occurring in the 90 days following inclusion in patients in the intervention group for whom PE was ruled out according to the 4PEPS strategy and who were not treated with anticoagulants.
Rate of thromboembolic events occurring in the 90 days following inclusion in patients for whom PE was ruled out in both groups | 90 days
  The second secondary objective is to demonstrate that the 4PEPS strategy (intervention group) is not inferior to current practices (control group) as regards the risk of false-negative diagnosis.
  The false-negative rate will be defined as the rate of thromboembolic events occurring in the 90 days following inclusion in patients for whom PE was ruled out and who were not treated with anticoagulants.
Rate of D-dimer measurement | up to 72 hours following inclusion
  The third secondary objective is to to evaluate and compare to usual practice the impact of the 4PEPS strategy as regards the rate of D-dimer measurement.
Length of stay in ED | Up to Emergency Department discharge (assessed up to 48 hours)
  The fourth secondary objective is to evaluate and compare to usual practice the impact of the 4PEPS strategy as regards the length of time spent in the emergency department by patients with suspected PE.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Marie ROY, MD, PhD, Principal Investigator — University Hospital, Angers
Locations (23):
- Belgium (2):
  - Cliniques Bruxelles, Brussels
  - CHU Liège, Liège
- France (21):
  - CH Agen, Agen
  - CHU Angers, Angers
  - CH Argenteuil, Argenteuil
  - CH Arpajon, Arpajon
  - AP HP Clamart, Clamart
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - CH La Rochelle, La Rochelle
  - CH Versailles, Le Chesnay
  - CHU Limoges, Limoges
  - CHU Lyon, Lyon
  - CHR Metz Thionville, Metz
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - GH Paris, Paris
  - CHU Poitiers, Poitiers
  - CH Rochefort, Rochefort
  - CHU Rouen, Rouen
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours
  - CH Troyes, Troyes

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared at a later date upon request (e.g., the CRF to allow a collaborator to select the data they wish to access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the study investigator, based on a protocol provided by the requester, after verification of the obtaining of regulatory approvals, including the favorable opinion of an ethics committee.
Supporting Information: Study Protocol
Time Frame: The study protocol is already published and available (doi: 10.3390/diagnostics12123101). The data will be shared after signing a negotiated data transfer agreement ( data access agreement), for the duration specified in the agreement.
Access Criteria: The data will be made available via secure transfer (sharing platform approved by the university hospital: BlueFiles or Oodrive).

REFERENCES:
- [Background] Roy PM, Friou E, Germeau B, Douillet D, Kline JA, Righini M, Le Gal G, Moumneh T, Penaloza A. Derivation and Validation of a 4-Level Clinical Pretest Probability Score for Suspected Pulmonary Embolism to Safely Decrease Imaging Testing. JAMA Cardiol. 2021 Jun 1;6(6):669-677. doi: 10.1001/jamacardio.2021.0064. PMID 33656522
- [Background] Roy PM, Durieux P, Gillaizeau F, Legall C, Armand-Perroux A, Martino L, Hachelaf M, Dubart AE, Schmidt J, Cristiano M, Chretien JM, Perrier A, Meyer G. A computerized handheld decision-support system to improve pulmonary embolism diagnosis: a randomized trial. Ann Intern Med. 2009 Nov 17;151(10):677-86. doi: 10.7326/0003-4819-151-10-200911170-00003. PMID 19920268
- [Background] Roy PM, Moumneh T, Penaloza A, Schmidt J, Charpentier S, Joly LM, Riou J, Douillet D. Diagnostic Strategy for Suspected Pulmonary Embolism in Emergency Departments Based on the 4-Level Pulmonary Embolism Clinical Probability Score: Study Protocol of SPEED&PEPS Trial. Diagnostics (Basel). 2022 Dec 9;12(12):3101. doi: 10.3390/diagnostics12123101. PMID 36553108